CLINICAL TRIAL: NCT05772117
Title: A Randomized Controlled Trial Evaluating a Theory-based Online Intervention Via Fully Automated Chatbot in Increasing Pneumococcal Vaccination Among Community Dwelling Individuals Aged ≥65 Years
Brief Title: A RCT Evaluating an Online Intervention in Increasing Pneumococcal Vaccination Among Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Zixin Wang, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20190972
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Vaccination Refusal
MeSH Terms: conditions — Vaccination Refusal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants receive Chatbot-delivered interventions tailored to their stage of change regarding PV uptake in a conversational way at Month 0, 1, 2, and 3.
  Interventions: Behavioral: Chatbot-delivered interventions tailored to stage of changes
- Control (Active Comparator): Participants receive Chatbot-delivered general information related to PV at Month 0, 1, 2, and 3.
  Interventions: Behavioral: Chatbot-delivered standard interventions

INTERVENTIONS:
Behavioral: Chatbot-delivered interventions tailored to stage of changes — Participants receive Chatbot-delivered interventions tailored to their stage of change regarding PV uptake in a conversational way at Month 0, 1, 2, and 3.
  Arms: Intervention
Behavioral: Chatbot-delivered standard interventions — Participants receive Chatbot-delivered general information related to PV at Month 0, 1, 2, and 3.
  Arms: Control

SUMMARY:
To evaluate the relative efficacy of an online intervention based on the Trans-theoretical Model delivered by a fully-automated Chatbot with natural language processing functions versus a control in promoting pneumococcal vaccination uptake among Hong Kong people aged ≥65 years. A total of 374 participants will be randomized evenly to either the intervention group or the control group. Participants in the intervention group will receive Chatbot-delivered interventions tailored to their stage of change regarding PV uptake in a conversational way at Month 0, 1, 2, and 3. Participants in the control group will receive Chatbot-delivered general information related to PV at Month 0, 1, 2, and 3. All participants will be followed up 6 and 12 months after completion of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥65 years
* having Hong Kong ID
* Chinese speaking
* have not received any penumococcal vaccination
* willing to be followed up by telephone
* having a smartphone
* able to send and read text/voice messages via smartphone.

Exclusion Criteria:

* blindness or deafness
* not able to communicate with others effectively
* with known contradictions of pneumococcal vaccination
* having been diagnosed with major psychiatric illness
* scored ≤16 in the validated telephone version of the Cantonese Mini-mental State Examination (T-CMMSE).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 374 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Pneumococcal vaccination uptake | 12 months
  Self-reported uptake of pneumococcal vaccination within the 12-month follow-up period

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Health Behaviours Research, the Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang Z, Chen S, Poon J, Han SC, Ye D, Yu FY, Fang Y, Ni Z, Wong MCS, Mo PKH. A Hybrid Chatbot to Promote Pneumococcal Vaccination Among Older Adults: A Randomized Clinical Trial. JAMA Netw Open. 2025 Oct 1;8(10):e2535813. doi: 10.1001/jamanetworkopen.2025.35813. PMID 41060654